CLINICAL TRIAL: NCT00767598
Title: The Effect of CYP3A Genetic Polymorphism on the Pharmacokinetics of Phosphodiesterase type5 Inhibitors(PDE5I) in Male Subjects
Brief Title: The Effect of CYP3A Genetic Polymorphism on the Pharmacokinetics of Phosphodiesterase type5 Inhibitors in Male Subjects
Acronym: CYP3APDE5I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Department of Pharmacology and PharmacoGenomics Research Center, Inje University College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 07-109
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-07

CONDITIONS: Pharmacokinetics of Three PDE5Is; Healthy Subjects; Genetic Polymorphic CYP3A5
Keywords: CYP3A5; sildenafil; udenafil; vardenafil
MeSH Terms: interventions — Phosphodiesterase 5 Inhibitors; Vardenafil Dihydrochloride; Sildenafil Citrate; udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Vardenafil
  Interventions: Drug: phosphodiesterase type 5 inhibitor
- B (Active Comparator): Sildenafil
  Interventions: Drug: phosphodiesterase type 5 inhibitor
- C (Active Comparator): Udenafil
  Interventions: Drug: phosphodiesterase type 5 inhibitor

INTERVENTIONS:
Drug: phosphodiesterase type 5 inhibitor — single oral administration of 20mg vardenafil
  Other Names: vardenafil
  Arms: A
Drug: phosphodiesterase type 5 inhibitor — single oral administration of 100mg sildenafil
  Other Names: sildenafil
  Arms: B
Drug: phosphodiesterase type 5 inhibitor — single oral administration of 200mg udenafil
  Other Names: udenafil
  Arms: C

SUMMARY:
In order to evaluate the effect of CYP3A5*3 allele on the pharmacokinetics of sildenafil, udenafil, and vardenafil, the clinical trial using a single oral dose was conducted in Korean healthy male subjects whose genotype of CYP3A5 had been determined.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the different effect of the CYP3A5 genotype on the pharmacokinetics(PK) of sildenafil, udenafil, and vardenafil in healthy male subjects. Twenty one healthy male subjects with CYP3A5*1/*1, *1/*3, or *3/*3 were enrolled. An open-label 3-way crossover study was performed with a week washout. A single oral dose of PDE5I (100 mg sildenafil; 200 mg udenafil; 20 mg vardenafil) was administered, respectively. After a single oral dose of phosphodiesterase type 5 inhibitor (PDE5I), plasma levels of the parent and the major metabolite were measured up to 24 or 48 h.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject whose CYP3A5 genotype was determined

Exclusion Criteria:

* Subject whose CYP3A5 genotype was not determined

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-12; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Cmax, AUC | upto 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, Principal Investigator — Inje University